CLINICAL TRIAL: NCT06932315
Title: A Study to Evaluate the Safety, Tolerability and Dose-Response Relationship of HRS-9190 in Healthy Adults
Brief Title: A Study to Evaluate the Safety, Tolerability and Dose-Response Relationship of HRS-9190 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-9190-101
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Skeletal Muscle Relaxation
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-9190 Experimental Group (Experimental)
  Interventions: Drug: HRS-9190 for Injection

INTERVENTIONS:
Drug: HRS-9190 for Injection — Subject will receive the HRS-9190 injection at different dose levels.

SUMMARY:
This is a single-center, open-label and dose-escalation study to evaluate the safety, tolerability and dose-response relationship of HRS-9190 in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects aged 18 to 45 years (inclusive).
2. Subjects must have no pregnancy plans for the next three months and agree to use highly effective contraception throughout the trial period.
3. Capable of understanding the study requirements and willing to provide written informed consent.

Exclusion Criteria:

1. Presence of any clinically significant condition that could interfere with trial participation.
2. History or current diagnosis of neuromuscular disorders.
3. Major surgery within 6 months pre-screening, or planned surgical procedures during the study.
4. Vaccination received within 1 month prior to screening or planned vaccination during the trial period.
5. Participation in another investigational drug trial within 3 months pre-screening.
6. Clinically significant abnormalities in screening/baseline physical examinations.
7. Positive alcohol breath test at screening.
8. Pregnancy or lactation status (for female subjects).
9. Investigator-determined unsuitability for study participation or predicted protocol non-compliance.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | From the ICF signing date to Day 7.

SECONDARY OUTCOMES:
The maximum observed concentration of HRS-9190 (Cmax) | 0 hour to 1.5 hours after administration.
Time to Cmax of HRS-9190 (Tmax) | 0 hour to 1.5 hours after administration.
Terminal elimination half-life of HRS-9190 (t1/2) | 0 hour to 1.5 hours after administration.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided